CLINICAL TRIAL: NCT01172457
Title: A Randomized, Double-Blind Study to Evaluate the Effect of Epiduroscopy and Ozone Therapy in Patients With Failed Back Surgery Syndrome
Brief Title: The Effect of Epiduroscopy and Ozone Therapy in Patients With Failed Back Surgery Syndrome
Acronym: Epiduroscopy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Neuton Magalhaes, MD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Epiduroscopy trial
Record Dates: First submitted 2010-07-28; First posted 2010-07-29 (Estimated); Last update posted 2013-08-30 (Estimated); Status verified 2013-08

CONDITIONS: Low Back Pain; Failed Back Surgery Syndrome
Keywords: low back pain; failed back surgery syndrome (FBSS); epidural fibrosis; ozone therapy; oxygen therapy; epiduroscopy; spinal endoscopy
MeSH Terms: conditions — Low Back Pain; Failed Back Surgery Syndrome | interventions — Oxygen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Epiduroscopy with ozone therapy (Active Comparator): Patients in this group will receive 30 mL of ozone at a concentration of 30 mcg / ml by epiduroscopy.
  Interventions: Procedure: Epiduroscopy with ozone therapy
- Epiduroscopy with oxygen therapy (Placebo Comparator): Patients in this group will receive 30 mL of oxygen by epiduroscopy.
  Interventions: Procedure: Epiduroscopy with oxygen therapy

INTERVENTIONS:
Procedure: Epiduroscopy with oxygen therapy — Patients in this group will receive 30 mL of oxygen by epiduroscopy.
  Arms: Epiduroscopy with oxygen therapy
Procedure: Epiduroscopy with ozone therapy — Patients in this group will receive 30 mL of ozone at a concentration of 30 mcg / ml by epiduroscopy.
  Arms: Epiduroscopy with ozone therapy

SUMMARY:
The aim of this study is to assess the efficacy and safety of ozone therapy (vs. placebo) applied into the epidural space through epiduroscopy in Patients with Failed Back Surgery Syndrome. It´s a Prospective, double blind, randomized study. The investigators will study 30 patients of both sexes between 18 and 70 years with chronic back pain after lumbar spine surgery for more than six months. The patients will receive the ozone gas or placebo (oxygen) in the lumbar epidural space, using a spinal endoscope inserted through the sacral hiatus by local anesthesia or sedation. The patients will be evaluated before the procedure, with 30 days, with 3, 6 and 12 months after intervention. This will be run by a researcher who will have no knowledge of the gas (oxygen or ozone) to be injected into the lumbar epidural space with the aid of an epiduroscopic. Will be applied before and after the procedure, pain scales (VAS, McGill, Neuropathic Pain 4, Neuropathic Pain Symptom Inventory), quality of life scale (WHOQOL), functional scales of pain disability (Roland Morris and Oswestry Disabilities Scales). Only one researcher will keep the data confidential until the end of the study.

DETAILED DESCRIPTION:
Although surgical discectomy for disc herniation produces better short-term pain relief than conservative therapy, there is no convincing evidence for the long-term (10 years) advantage of surgery. Between 40% and 80% of patients undergoing back surgery continue to experience persistent pain, a condition called Failed Back Surgery Syndrome (FBSS). The symptoms of FBSS are of persistent or recurring low back pain and / or leg pain after one or more spinal operations. The precise cause of the pain can be difficult to determine due to the complex interaction of biological and psychosocial factors. Possible organic causes of FBSS include epidural fibrosis, arachnoiditis, mechanical factors, pressure induced changes in the nerve root, structural changes in the vertebral column, and lumbar degenerative disease. With a second surgical intervention for fibrosis, there is a 65-70% failure rate, with 15-20% of the patients reporting worsening of symptoms. Thus, repeated surgery tends to yield poorer results.

The ozone therapy has emerged as an option or additional treatment for these patients, mostly in Europe. Despite of its wide use to treat a variety of conditions, ozone therapy is still unknown to most physicians. Ozone (O3) is an allotropic form of oxygen, primarily known for its ecological properties, industrial applications, but also by its therapeutic effects. Some questions persist concerning its potential toxicity as an oxidant agent versus the reported clinical efficacy. Several mechanisms of action have been proposed to explain the efficacy of the ozone therapy: analgesic, anti-inflammatory and oxidant action on proteoglycan (e.g. in the nucleus pulpous). Ozone is administered in the form of an oxygen-ozone gas mixture at nontoxic concentrations varying from 1 to 40 µg of ozone per milliliter of oxygen by various percutaneous methods for treatment of low back pain. However, still no well-designed studies that allow conclusions about the safety and efficacy of ozone in the treatment of low back pain.

Spinal endoscopy, or "epiduroscopy", is the examination of the epidural space by a minimally invasive technique that allows the diagnosis and treatment of chronic back pain and radiculopathy. The therapeutic potential of epiduroscopy and adhesiolysis, a minimally invasive but potentially useful treatment modality in the management of refractory radiculopathy, emerged during the 1990s.

Epiduroscopy is carried out under local anesthesia with the patient awake, thus avoiding potential unrecognized pressure effects in the epidural canal. Light intravenous sedation and analgesia may be required to ensure full patient cooperation while maintaining verbal contact. The patient is positioned prone with a pillow under his/her hips. The procedure is carried out under aseptic conditions with antibiotic prophylaxis and requires the use of an imagine intensifier. Sacrococcygeal ligament puncture is made with a 17g Tuohy needle and followed by a caudal epidurogram to confirm needle placement. A Seldinger technique is then used to place an introducer sheath in the sacral epidural canal. A 0.9mm fiber optic scope is placed with its tip and the end of a steerable video guided catheter.

The Video Guided Catheter and endoscope are then advanced via the introducer into epidural space. Slow irrigation with saline allows visualization of epidural space by gentle distension. Adhesiolysis can be carried out under direct vision by blunt dissection of the adhesions using the tip of the video guided catheter. Blunt dissection coupled with hydrostatic distension of the epidural space thus creates a pocket through which injected drug can access symptomatic nerve roots.

Several drugs have been used within the epidural space through the spinal endoscopy including steroid, local anesthetic, hyaluronidase, saline solution, clonidine and ozone most recently. Blind epidural injections of these therapeutic substances can, in some patients; fail to flow towards a symptomatic root due to obstruction by epidural fibrosis. Such patients may, therefore, benefit more from epidural injection if flow of inject towards the symptomatic root is facilitated following endoscopic division of epidural adhesions.

Thus, the investigators find this model of pain would be appropriate to evaluate the effects of ozone in treatment for the lumbar pain by comparison with a placebo, using the epiduroscopy to apply it.

ELIGIBILITY:
Inclusion Criteria:

* Sciatic pain of 5 or more on Visual Analogue Scale
* Previous lumbar spine surgery
* More than six months into group interdisciplinary pain with pain refractory to medical treatment
* Patients with FBSS of the nonsurgical etiology
* Patients without labor dispute ort secondary gain

Exclusion Criteria:

* Inability to fill out questionnaires (VAS, Roland Morris, WHOQOL, OSWESTRY DISABILITY SCALE, f. ex.)
* Presence of other spinal pathology
* Allergy to ozone
* Treatment with oral anticoagulants
* Hyperthyroidism
* Diabetic neuropathy
* favism (Significant glucose-6-phosphate-dehydrogenase deficit)and hyperthyroidism that are contra-indications for ozone therapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-05; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of ozone versus placebo (oxygen) applied into the epidural space of patients with Failed Back Surgery Syndrome (FBSS) through epiduroscopy. | up to 01 year
  The pain intensity is measured by visual analog pain scale - VAS

SECONDARY OUTCOMES:
To evaluate the psychological aspects. | up to 01 year
  To evaluate the effects of ozone applied into the epidural space of patients with Failed Back Surgery Syndrome (FBSS) through epiduroscopy about the psychological aspects. The investigators are using the Beck Depression Inventory.
The quality of life. | up to 01 year
  To evaluate the effects of ozone applied into the epidural space of patients with chronic pain syndrome post-laminectomy through epiduroscopy about the quality of life using the WHOQOL questionaire.
To evaluate the physical capacity | up to 01 year
  To evaluate the effects of ozone applied into the epidural space of patients with chronic pain syndrome post-laminectomy through epiduroscopy about physical capacity. The investigators are using the Oswestry Disability Index.
To evaluate the use of analgesic medications | up to 01 year
  The researchers will evaluate the amount of analgesic medications used during the monitoring period.
To evaluate the rate of side effects or complications | up to 01 year
  The side effects or adverse effects will be assessed according to Common Terminology Criteria for Adverse Effect 4.0. In case of complications, will be recorded and analyzed.

CONTACTS AND LOCATIONS:
Locations (1):
- University of São Paulo Medical School, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Gillespie G, MacKenzie P. Epiduroscopy--a review. Scott Med J. 2004 Aug;49(3):79-81. doi: 10.1177/003693300404900301. No abstract available. PMID 15462218
- [Background] Geurts JW, Kallewaard JW, Richardson J, Groen GJ. Targeted methylprednisolone acetate/hyaluronidase/clonidine injection after diagnostic epiduroscopy for chronic sciatica: a prospective, 1-year follow-up study. Reg Anesth Pain Med. 2002 Jul-Aug;27(4):343-52. doi: 10.1053/rapm.2002.27175. PMID 12132057
- [Background] Manchikanti L, Pampati V, Cash KA. Protocol for evaluation of the comparative effectiveness of percutaneous adhesiolysis and caudal epidural steroid injections in low back and/or lower extremity pain without post surgery syndrome or spinal stenosis. Pain Physician. 2010 Mar-Apr;13(2):E91-E110. PMID 20309389
- [Background] Manchikanti L, Singh V, Cash KA, Pampati V, Datta S. A comparative effectiveness evaluation of percutaneous adhesiolysis and epidural steroid injections in managing lumbar post surgery syndrome: a randomized, equivalence controlled trial. Pain Physician. 2009 Nov-Dec;12(6):E355-68. PMID 19935992
- [Background] Manchikanti L, Boswell MV, Datta S, Fellows B, Abdi S, Singh V, Benyamin RM, Falco FJ, Helm S, Hayek SM, Smith HS; ASIPP. Comprehensive review of therapeutic interventions in managing chronic spinal pain. Pain Physician. 2009 Jul-Aug;12(4):E123-98. PMID 19668281
- [Background] Hayek SM, Helm S, Benyamin RM, Singh V, Bryce DA, Smith HS. Effectiveness of spinal endoscopic adhesiolysis in post lumbar surgery syndrome: a systematic review. Pain Physician. 2009 Mar-Apr;12(2):419-35. PMID 19305488
- [Background] Epter RS, Helm S 2nd, Hayek SM, Benyamin RM, Smith HS, Abdi S. Systematic review of percutaneous adhesiolysis and management of chronic low back pain in post lumbar surgery syndrome. Pain Physician. 2009 Mar-Apr;12(2):361-78. PMID 19305485
- [Background] Sakai T, Aoki H, Hojo M, Takada M, Murata H, Sumikawa K. Adhesiolysis and targeted steroid/local anesthetic injection during epiduroscopy alleviates pain and reduces sensory nerve dysfunction in patients with chronic sciatica. J Anesth. 2008;22(3):242-7. doi: 10.1007/s00540-008-0616-4. Epub 2008 Aug 7. PMID 18685930
- [Background] Racz GB, Heavner JE, Trescot A. Percutaneous lysis of epidural adhesions--evidence for safety and efficacy. Pain Pract. 2008 Jul-Aug;8(4):277-86. doi: 10.1111/j.1533-2500.2008.00203.x. Epub 2008 May 23. PMID 18503627
- [Background] Boswell MV, Trescot AM, Datta S, Schultz DM, Hansen HC, Abdi S, Sehgal N, Shah RV, Singh V, Benyamin RM, Patel VB, Buenaventura RM, Colson JD, Cordner HJ, Epter RS, Jasper JF, Dunbar EE, Atluri SL, Bowman RC, Deer TR, Swicegood JR, Staats PS, Smith HS, Burton AW, Kloth DS, Giordano J, Manchikanti L; American Society of Interventional Pain Physicians. Interventional techniques: evidence-based practice guidelines in the management of chronic spinal pain. Pain Physician. 2007 Jan;10(1):7-111. PMID 17256025
- [Background] Manchikanti L, Pampati V, Fellows B, Rivera JJ, Damron KS, Beyer C, Cash KA. Effectiveness of percutaneous adhesiolysis with hypertonic saline neurolysis in refractory spinal stenosis. Pain Physician. 2001 Oct;4(4):366-73. PMID 16902683
- [Background] Mavrocordatos P, Cahana A. Minimally invasive procedures for the treatment of failed back surgery syndrome. Adv Tech Stand Neurosurg. 2006;31:221-52. doi: 10.1007/3-211-32234-5_5. PMID 16768306
- [Background] Steppan J, Meaders T, Muto M, Murphy KJ. A metaanalysis of the effectiveness and safety of ozone treatments for herniated lumbar discs. J Vasc Interv Radiol. 2010 Apr;21(4):534-48. doi: 10.1016/j.jvir.2009.12.393. Epub 2010 Feb 25. PMID 20188591
- [Background] Das G, Ray S, Ishwarari S, Roy M, Ghosh P. Ozone nucleolysis for management of pain and disability in prolapsed lumber intervertebral disc. A prospective cohort study. Interv Neuroradiol. 2009 Sep;15(3):330-4. doi: 10.1177/159101990901500311. Epub 2009 Nov 4. PMID 20465917
- [Background] Paoloni M, Di Sante L, Cacchio A, Apuzzo D, Marotta S, Razzano M, Franzini M, Santilli V. Intramuscular oxygen-ozone therapy in the treatment of acute back pain with lumbar disc herniation: a multicenter, randomized, double-blind, clinical trial of active and simulated lumbar paravertebral injection. Spine (Phila Pa 1976). 2009 Jun 1;34(13):1337-44. doi: 10.1097/BRS.0b013e3181a3c18d. PMID 19478653
- [Background] Staal JB, de Bie RA, de Vet HC, Hildebrandt J, Nelemans P. Injection therapy for subacute and chronic low back pain: an updated Cochrane review. Spine (Phila Pa 1976). 2009 Jan 1;34(1):49-59. doi: 10.1097/BRS.0b013e3181909558. PMID 19127161
- [Background] Muto M, Ambrosanio G, Guarnieri G, Capobianco E, Piccolo G, Annunziata G, Rotondo A. Low back pain and sciatica: treatment with intradiscal-intraforaminal O(2)-O (3) injection. Our experience. Radiol Med. 2008 Aug;113(5):695-706. doi: 10.1007/s11547-008-0302-5. Epub 2008 Jul 1. English, Italian. PMID 18594765
- [Background] Oder B, Loewe M, Reisegger M, Lang W, Ilias W, Thurnher SA. CT-guided ozone/steroid therapy for the treatment of degenerative spinal disease--effect of age, gender, disc pathology and multi-segmental changes. Neuroradiology. 2008 Sep;50(9):777-85. doi: 10.1007/s00234-008-0398-2. Epub 2008 May 16. PMID 18483728
- [Background] Gallucci M, Limbucci N, Zugaro L, Barile A, Stavroulis E, Ricci A, Galzio R, Masciocchi C. Sciatica: treatment with intradiscal and intraforaminal injections of steroid and oxygen-ozone versus steroid only. Radiology. 2007 Mar;242(3):907-13. doi: 10.1148/radiol.2423051934. Epub 2007 Jan 5. PMID 17209164
- [Background] Bertoli AM, Alarcon GS. Ozone therapy and lower back pain. AJNR Am J Neuroradiol. 2006 Mar;27(3):471; author reply 471. No abstract available. PMID 16551979
- [Background] Bonetti M, Fontana A, Cotticelli B, Volta GD, Guindani M, Leonardi M. Intraforaminal O(2)-O(3) versus periradicular steroidal infiltrations in lower back pain: randomized controlled study. AJNR Am J Neuroradiol. 2005 May;26(5):996-1000. PMID 15891150
- [Background] Bonetti M, Fontana A, Albertini F. CT-guided oxygen-ozone treatment for first degree spondylolisthesis and spondylolysis. Acta Neurochir Suppl. 2005;92:87-92. doi: 10.1007/3-211-27458-8_19. PMID 15830975
- [Background] Muto M, Andreula C, Leonardi M. Treatment of herniated lumbar disc by intradiscal and intraforaminal oxygen-ozone (O2-O3) injection. J Neuroradiol. 2004 Jun;31(3):183-9. doi: 10.1016/s0150-9861(04)96989-1. PMID 15356443
- [Result] Fai KR, Engleback M, Norman JB, Griffiths R. Interlaminar approach for epiduroscopy in patients with failed back surgery syndrome. Br J Anaesth. 2009 Feb;102(2):280; author reply 280-1. doi: 10.1093/bja/aen371. No abstract available. PMID 19151054
- See also: Related Info — http://www.aboz.com.br